CLINICAL TRIAL: NCT05577013
Title: Combined Effects of Kinesiotaping and Motor Relearning Program on Upper Limb Motor Function After Stroke
Brief Title: Kinesio Taping Versus Motor Relearning Program for Upper Limb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-01043 Rabia
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Kinesiotaping and motor relearning program group (Experimental): The experimental group will receive kinesiotaping; Instructions before applying kinesiotape
  * Patients' skin must be clean, free of dirt, oil or sweat.
  * Long hair must be removed for proper adhesion to the skin.
  * Leave the tape upstretched 2-3 cm at start and end point of tape over the skin
  Interventions: Other: kinesiotaping
- motor relearning program group (Active Comparator): The control group will receive motor relearning programme exercises for 40 minutes.
  1. Hitting a target on table from flexed elbow to extension of elbow
  2. Hitting a target on front of table with shoulder flexion (reaching fwd)
  3. Hitting a target on table with wrist extension
  4. Pronation to supination while holding a bottle of water.
  5. Rolling ball on table in forward, backward and sideways
  6. Holding polystyrene cup and placing it on other side
  7. Picking up blocks and placing them to other side
  8. Holding polystyrene cup and placing them above and below level of sitting to front and sideways
  9. Holding polystyrene cup and placing them above and below level of standing to front and sideways
  10. pick small objects from one container to another
  Interventions: Other: motor relearning program

INTERVENTIONS:
Other: kinesiotaping — It will be applied by kinesiotape certified physiotherapist on tendons in the direction of extensor muscle to facilitate range of motion by stretching 50%. At first it will be applied on extensor pollicis longus and extensor pollicis brevis muscles of hand, extensor digitorum and extensor indicis of last 4 fingers of hand. Triceps brachii in arm and Supraspinatus and Infraspinatus muscles to stabilize the gelnohumeral joint
  Arms: (Kinesiotaping and motor relearning program group
Other: motor relearning program — Stacking up blocks Stacking up polystyrene cups Folding piece of cloth Using cutlery Pouring water into glass Closing/opening lid of bottles turning the pages of books or newspaper writing on paper Squeezing of ball Coloring in different shapes
  Arms: motor relearning program group

SUMMARY:
Stroke is described as rapidly developing clinical findings of localized or generalized impairment to cerebral function, with symptoms lasting 24 hours or longer, or leading to death, with no evident cause other than a vascular origin.

Stroke is a prevalent and debilitating illness that affects people all around the world. Stroke is the second or third largest cause of mortality in adults, as well as one of the primary causes of adult disability. Because the majority of stroke patients survive the initial illness, the long-term impacts on patients and their families have the greatest influence on health. Kinesiotaping is a revolutionary rehabilitation procedure. It's most typically used to treat sports injuries, however, it is progressively becoming effective in overcoming other abnormalities. Kinesio Tex tape brand is a flexible, thin, porous cotton fabric with an adhesive backing manufactured by Dr. Kenzo Kase. It provides cutaneous stimulation which facilitates or limit movement, aids in the reduction of edema, reduces pain and correct joint positions for easing muscle spasms.

ELIGIBILITY:
Inclusion Criteria:

* male and female of age 18 -60 years
* patients with post stroke duration of >6 months
* both ischemic and hemorrhagic stroke
* modified ashworth scale of spasticity < 3
* muscle power by manual muscle testing (MMT) ≥ 2
* no cognitive impairments by mini mental state examination (MMSE) > 24
* cortical skin sensitivity preserved (two point discrimination, barognosis, fine and crude touch)

Exclusion Criteria:

* Participants failing to fall in this category would be excluded from the study.
* being hospitalized due to any reason other than stroke
* being subjected to treatment with botulinum toxin for <1 year
* any other condition which affects the upper extremity
* contraindications for the application of Kinesio Taping: open wounds, skin infections such as cellulitis, allergies, skin xerosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Fugel Meyer assessment scale for upper limb | week 8
  An assessment scale for post stroke hemiplegic patients and is performance-based impairment index. This scale is having 5 domains namely Motor functioning, Sensory Functioning, Balance, Joint Range of Motion and Joint pain. I divided the motor functioning for upper extremity into 0 to 66 points and evaluates mobility, speed and coordination
Functionality of Upper Limb | week 8
  Upper Limb functionality is assessed by an instrument that consists of 20 items divided into 13 items that evaluate the movement patterns of the upper limb with a score from 0 (paralysis) to 5 (performs the typical movement pattern compared to the unaffected side)
Box and Block Test (BBT) | week 8
  his test is used to evaluate the manual dexterity of post stroke patients. BBT is composed of wooden box with two equal compartments having 150 boxes in one compartment and patient is asked to move the boxes from one compartment to another within 60 seconds. Before starting the test an extra 15 seconds time is given to the patient for familiarization with the test. First the patient performed the activity with the healthy arm and then with the affected arm. Scoring is done on the basis of the number of boxes transferred from one compartment to another within 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Afridi, PhD, Principal Investigator — Riphah International University
Locations (1):
- Rehman Medical Institute, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No